CLINICAL TRIAL: NCT03252145
Title: Treatment of Breast Cancer-related Lymphedema With a Negative Pressure Device: A Feasibility Study
Brief Title: Treatment of Breast Cancer-related Lymphedema With a Negative Pressure Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Foundation for Physical Therapy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P0518095; NCI-2018-00009 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); 16802 (Other: University of California, San Francisco)
Record Dates: First submitted 2017-08-10; First posted 2017-08-17 (Actual); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Lymphedema, Secondary; Lymphedema of Upper Limb
MeSH Terms: conditions — Lymphedema; Neoplasm Metastasis | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Negative Pressure (Experimental): PhysioTouch (negative pressure massage) treatment 3 times a week for 4 weeks to the lymphedematous upper limb
  Interventions: Device: PhysioTouch
- Manual Lymph Drainage (Active Comparator): Manual lymph drainage (MLD) treatment 3 times a week for 4 weeks to the lymphedematous upper limb
  Interventions: Other: Manual Lymph Drainage (MLD)

INTERVENTIONS:
Device: PhysioTouch — The PhysioTouch is a hand-held device that administers negative pressure under the treatment head, and gently pulls the underlying skin and subcutaneous tissue into the suction cup. This suction produces a stretch to the skin and in the subcutaneous tissue space. This action is thought to facilitate lymphatic flow from the interstitium into the lymphatic vessels, and mobilizes the superficial fascia.
  Arms: Negative Pressure
Other: Manual Lymph Drainage (MLD) — MLD is a practitioner-applied manual massage technique designed to decrease limb volume in patients with lymphedema by enhancing movement of lymph fluid, resulting in reductions in interstitial fluid.
  Arms: Manual Lymph Drainage

SUMMARY:
This study will be a 4 to 6 week randomized, controlled, assessor blinded, trial comparing a negative pressure massage device (intervention group), to the standard manual lymph drainage massage (control group), in breast cancer patients with chronic upper extremity lymphedema.

DETAILED DESCRIPTION:
Lymphedema (LE) is a protein-rich interstitial swelling caused by reduced lymph transport secondary to lymphatic system damage from cancer treatments. 1 in 5 women will develop LE following breast cancer treatment. These women have greater restrictions in activity and poorer quality of life (QOL) and are more prone to cellulitis than women without LE. LE is incurable and progressive. Persistent lymph stasis creates a condition of chronic inflammation that contributes to fibrosis and fatty deposition in the subcutis of the affected limb. The fibro-adipose changes associated with chronic LE make it less responsive to treatments that primarily target limb volume. Treatments are needed that can improve these skin and subcutaneous tissues changes, as well as reduce limb volume.

This 4 to 6 week randomized controlled pilot feasibility study will enroll 80 women with chronic arm LE, and will evaluate a novel negative pressure massage device that mobilizes skin and subcutaneous tissue. This negative pressure treatment provides vertical (lifting) and horizontal stretching of the skin and underlying fascial structures, which increases the subcutaneous space for lymphatic circulation, improves lymph flow, and has the potential to decrease fibrosis. This treatment will be compared to the standard of care massage: manual lymphatic drainage. Women will be randomly assigned to either the negative pressure massage device (intervention group), to the standard manual lymph drainage massage (control group)

Objectives: To evaluate recruitment and retention rates; to determine rates of adverse events; and to determine effect sizes for limb volume, tissue induration; and patient reported outcomes of arm function, QOL, and body image in response to treatment

ELIGIBILITY:
INCLUSION CRITERIA:

To be included women must be:

Be over 18 years of age;

Have had cancer treatment that included a surgical procedure, radiation therapy (RT), and/or chemotherapy (CTX);

Have completed active cancer treatment at least 1 year prior to study enrollment;

Have been diagnosed with lymphedema (LE) at least one year prior to study enrollment;

Have arm lymphedema on one side only;

Have confirmed LE based on bioimpedance measurements with an L-Dex® score of >7.1 (note - this is very mild lymphedema);

Have stable arm LE. LE will be considered "stable" if during the 3 months prior to study enrollment there was no arm infection requiring antibiotics, no change in ability to perform activities of daily living related to LE, and no subjective report of significant persistent changes in limb volume;

Be mentally and physically able to participate in the study;

Be able to attend the sessions at the University of California, San Francisco (UCSF) Parnassus campus;

Read and understand English;

Be able to understand a written informed consent document and the willingness to sign it

EXCLUSION CRITERIA

Women cannot have:

* Bilateral upper extremity LE;
* Current infection or lymphangitis involving the affected arm;
* Current recurrence of their breast cancer (BC) (local or distant)
* Pre-existing LE prior to their BC diagnosis;
* A condition that precludes measurement of LE using Bioimpedance Spectroscopy (BIS), including pregnancy;
* Current venous thrombosis in either upper extremity or be on current anticoagulant therapy;
* Extremity edema due to heart failure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Betty Smoot, DPTSc, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lampinen R, Lee JQ, Leano J, Miaskowski C, Mastick J, Brinker L, Topp K, Smoot B. Treatment of Breast Cancer-Related Lymphedema Using Negative Pressure Massage: A Pilot Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 Aug;102(8):1465-1472.e2. doi: 10.1016/j.apmr.2021.03.022. Epub 2021 Apr 16. PMID 33872573

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a University of California, San Francisco 5-year cross-sectional study (CA187160). In addition, flyers were made available to participants at lymphedema and breast cancer conferences and patient symposia. Community collaborators (breast surgeons, lymphedema specialists, support group leaders) were also sent informational and recruitment materials related to the study.
Pre-assignment Details: Of the 130 who expressed interest in the study, only 28 met all inclusion criteria.
Period: Overall Study
Arm/Group | Manual Lymph Drainage | Negative Pressure
Started | 13 | 15
Completed | 11 | 13
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Complicating Disease | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Lymph Drainage | Negative Pressure | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 1 | 1 | 2
  40-49 years old | 1 | 1 | 2
  50-59 years old | 4 | 4 | 8
  60-69 years old | 5 | 3 | 8
  70-79 years old | 2 | 5 | 7
  80-89 years old | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 15 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 10 | 11 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rates
Description: The recruitment rate is defined as the number of women who were screened and then enrolled on the study divided by the the total number of women screened overall.
Time Frame: At 4 weeks
Measure: Number; unit: rate of recruitment
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 13 | 15
rate of recruitment | 32.5 | 37.5

2. Primary Outcome: Percentage of Participants Who Completed All Study Visits
Description: Retention rates for both arms of this study were evaluated. The numbers of women who completed the study will be recorded. Reasons for drop out will be ascertained.
Time Frame: At 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 13 | 15
percentage of participants | 84.6 | 86.7

3. Secondary Outcome: Mean Limb Volume
Description: Arm circumferential measurements of both limbs and hands were taken twice, using a spring-loaded tape measure. The hand was measured in two locations. Upper extremity measurements were taken at 10 centimeter (cm) intervals from the ulnar styloid of the wrist up to a total distance of 40 cm. Circumferences were measured using the procedures outlined by Cornish et al. Limb volume was calculated using the formula for volume of a truncated cone and reported in millilitre (ml)
Time Frame: At Baseline
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 13 | 15
ml | 383.32 (324.74) | 622.17 (396.39)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.096, t-test, 2 sided

4. Secondary Outcome: Mean Limb Volume
Description: as for outcome 3
Time Frame: At 4 weeks
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 13 | 15
ml | 352.66 (317.74) | 512.98 (332.77)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.206, t-test, 2 sided

5. Secondary Outcome: Mean Lymphedema Index (L-DEX®) Ratio Scores
Description: Bioimpedance spectroscopy (BIS) measurements were taken using a single channel BIS, tetrapolar device (LDex device, ImpediMed, San Diego, CA) to evaluate upper limb bioelectrical impedance. Impedance ratios (unaffected/affected limb) are calculated and converted to L-Dex ratio score. With development of lymphedema, impedance of extremity decreases and L-Dex ratio therefore increases. An L-Dex ratio score of 10 is equivalent to impedance ratio of 1.139 (which is = to 3 standard deviations (SD) from mean normative BIS data) for at-risk dominant arms & 1.066 for at-risk non-dominant arms, respectively. Each 1 standard unit in L-Dex is equivalent to impedance ratio of 0.03. Using this arbitrary scale relevant to normative standards, a patient is determined to have arm lymphedema if L-Dex ratio score exceeds 7.1, which is 2 SD above mean normative data for BIS impedance ratios. Higher L-Dex ratio score means higher impedance ratio between limbs, which means more volume in affected limb.
Time Frame: At Baseline
Population: The range of L-DEX ratio scores on our study at baseline were 0.1 - 74.20.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 13 | 15
score on a scale | 23.09 (20.87) | 34.16 (24.73)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.096, t-test, 2 sided

6. Secondary Outcome: Mean L-DEX® Scores
Description: as for outcome 5
Time Frame: At 4 weeks
Population: The range of L-DEX ratio scores on our study at 4 weeks were -2.85 - 77.50.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 13 | 15
score on a scale | 26.30 (22.23) | 30.09 (22.72)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.206, t-test, 2 sided

7. Secondary Outcome: Mean Skin Induration Score
Description: The SkinFibroMeter (Delfin Technologies, Finland) was used to measure tissue induration. The SkinFibroMeter consists of a 1 mm long indenter and a force sensor. The device is gently pressed against the skin. The indenter imposes a constant deformation when the reference plate is in full contact with the skin. The skin and the underlying superficial subcutis resist the deformation. Measurements will be taken bilaterally at 5 locations: the first dorsal web space; the medial forearm halfway between the ulnar styloid and medial epicondyle; the lateral forearm halfway between the radial styloid and the lateral epicondyle; the medial arm 3 inches proximal to the medial epicondyle; and the lateral arm 3 inches proximal to the lateral epicondyle. Five recordings were taken at each location and a mean score was calculated.The induration value in Newtons (N) is recorded.
Time Frame: At Baseline
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 13 | 15
Newtons | 0.077 (0.023) | 0.072 (0.021)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.552, t-test, 2 sided

8. Secondary Outcome: Mean Skin Induration Score
Description: as for outcome 7
Time Frame: At 4 weeks
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 13 | 15
Newtons | 0.069 (0.017) | 0.065 (0.017)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.498, t-test, 2 sided

9. Secondary Outcome: Mean Degrees of Shoulder Range of Motion
Description: Active shoulder flexion and abduction range of motion (ROM) was assessed, with patients supine, using a goniometer and standardized procedures reported by Norkin and White. Bilateral ROM was assessed. Two measurements will be taken for each motion and a mean obtained, for each, bilaterally. Findings are recorded in degrees.
Time Frame: At Baseline
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 13 | 15
degrees
  Affected arm | 167.5 (5.0) | 157.1 (34.0)
  Unaffected arm | 168.5 (6.9) | 163.7 (12.7)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Affected Arm Only; Test type: Other; p = 0.264, t-test, 2 sided
Statistical Analysis 2: Comparison: Manual Lymph Drainage vs Negative Pressure; Unaffected arm; Test type: Other; p = 0.224, t-test, 2 sided

10. Secondary Outcome: Mean Degrees of Shoulder Range of Motion
Description: as for outcome 9
Time Frame: At 4 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 13 | 15
degrees
  Affected arm | 170.5 (6.0) | 165.5 (9.5)
  Unaffected arm | 169.3 (7.5) | 164.6 (11.6)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Affected arm; Test type: Other; p = 0.125, t-test, 2 sided
Statistical Analysis 2: Comparison: Manual Lymph Drainage vs Negative Pressure; Unaffected arm; Test type: Other; p = 0.241, t-test, 2 sided

11. Secondary Outcome: Mean Grip Score
Description: Grip strength was assessed using a Jamar hydraulic hand dynamometer (Patterson Medical, Bolingbrook, IL). Patients will be tested in sitting with the feet flat on the floor, the arm at the side with the elbow flexed to 90 degrees. The patient was instructed to maximally squeeze the handle and hold for a count of 3. The peak-hold needle will automatically record the highest force exerted. Two trials for each extremity will be done and a mean grip score (in kilogram of force) calculated. A higher score indicates a greater grip strength.
Time Frame: At Baseline
Measure: Mean (Standard Deviation); unit: kilograms of force
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 13 | 15
kilograms of force
  Affected Arm | 24.0 (4.7) | 21.5 (6.4)
  Unaffected Arm | 25.7 (6.8) | 24.5 (4.3)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Affected Arm; Test type: Other; p = 0.261, t-test, 2 sided
Statistical Analysis 2: Comparison: Manual Lymph Drainage vs Negative Pressure; Unaffected Arm; Test type: Other; p = 0.597, t-test, 2 sided

12. Secondary Outcome: Mean Grip Score
Description: Grip strength was assessed using a Jamar hydraulic hand dynamometer (Patterson Medical, Bolingbrook, IL). Patients will be tested in sitting with the feet flat on the floor, the arm at the side with the elbow flexed to 90 degrees. The patient was instructed to maximally squeeze the handle and hold for a count of 3. The peak-hold needle will automatically record the highest force exerted. Two trials for each extremity will be done and a mean grip score (in kilograms of force) calculated. A higher score indicates a greater grip strength.
Time Frame: At 4 weeks
Measure: Mean (Standard Deviation); unit: kilograms of force
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 13 | 15
kilograms of force
  Affected arm | 26.4 (6.6) | 25.2 (4.1)
  Unaffected arm | 25.5 (6.1) | 22.6 (5.5)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Affected arm; Test type: Other; p = 0.596, t-test, 2 sided
Statistical Analysis 2: Comparison: Manual Lymph Drainage vs Negative Pressure; Unaffected arm; Test type: Other; p = 0.219, t-test, 2 sided

13. Secondary Outcome: Mean Karnofsky Performance Status (KPS) Score
Description: Participants rated their functional status using the single item KPS scale with a range from 0 (dead) to 100 (I feel normal; I have no complaints or symptoms), in increments of 10 (0,10,20, 30 , 40...). The lower the Karnofsky score, the worse the impairment.
Time Frame: At Baseline
Population: Only a subset of participants completed the questionnaire at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 12 | 13
score on a scale | 89.12 (13.79) | 88.18 (8.74)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.842, t-test, 2 sided

14. Secondary Outcome: Mean Karnofsky Performance Status (KPS) Score
Description: as for outcome 13
Time Frame: At 4 weeks
Population: Only a subset of participants completed the questionnaire at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 12 | 13
score on a scale | 91.8 (4.04) | 90.91 (9.44)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.772, t-test, 2 sided

15. Secondary Outcome: Mean Self-Administered Comorbidity Questionnaire (SCQ) Scores
Description: The SCQ consists of 13 common medical conditions that are simplified into language that could be understood without any prior medical knowledge. Patients were asked to indicate if they had the condition using a "yes/no" format. If they indicate that they had a condition, they are asked if they received treatment for it (yes/no; proxy for disease severity) and did it limit their activities (yes/no; indication of functional limitations). • For each condition, a patient can receive a maximum of 3 points. Because there are 13 defined medical conditions and 2 optional conditions, the maximum achievable total score is 45 points as all items were available for use.
Time Frame: At Baseline
Population: Only a subset of participants completed the questionnaire at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 12 | 11
score on a scale | 2.25 (2.09) | 3.42 (3.18)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.300, t-test, 2 sided

16. Secondary Outcome: Mean Self-Administered Comorbidity Questionnaire (SCQ) Scores
Description: as for outcome 15
Time Frame: 4 weeks
Population: Only a subset of participants completed the questionnaire at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 12 | 11
score on a scale | 2.25 (2.09) | 3.42 (3.18)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.300, t-test, 2 sided

17. Secondary Outcome: Mean Norman Questionnaire (NQ) Scores
Description: The NQ was originally developed and validated as a phone interview questionnaire to describe the signs and symptoms of breast cancer-related lymphoedema. Participants report subjective differences in the size of the hands, lower arms, and/or upper arms between their right and left sides. For each site difference, the reported score can range from 1 (very slight difference) to 3 (very noticeable difference). The total score can range from 1 (very slight difference at 1 site) to 9 (very noticeable difference at all 3 sites). Higher scores indicate a greater noticeable difference between the two arms
Time Frame: At Baseline
Population: Only a subset of participants completed the questionnaire at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 12 | 11
score on a scale | 3.83 (2.76) | 4.27 (2.20)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.679, t-test, 2 sided

18. Secondary Outcome: Mean Norman Questionnaire (NQ) Scores
Description: as for outcome 17
Time Frame: At 4 weeks
Population: Only a subset of participants completed the questionnaire at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 12 | 11
score on a scale | 2.75 (1.87) | 4.27 (2.61)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.120, t-test, 2 sided

19. Secondary Outcome: Mean Norman Questionnaire (NQ) Scores
Description: as for outcome 17
Time Frame: At 4 months
Population: Only a subset of participants completed the questionnaire at 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 7 | 9
score on a scale | 2.71 (1.89) | 4.56 (2.60)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.138, t-test, 2 sided

20. Secondary Outcome: Mean Disability of Arm, Shoulder, Hand Questionnaire (DASH) Scores
Description: The DASH is a 30-item self-report questionnaire measuring upper limb symptoms and ability to perform common functional activities in people with musculoskeletal disorders of the upper limb. The disability/symptom questions are scored 1 thru 5, with 1=being no difficulty and 5=being unable to perform. At least 27 of the 30 items must be completed for a scaled score to be calculated. The assigned values for all completed responses are simply summed and averaged, producing a raw score between 1 and 5. This value is then transformed to a score out of 100 to create a DASH disability/symptom score = [(sum of (n) responses) - 1] x 25, where n is equal to the number of completed responses. Each scaled score cut point is scored as 0 (no disability), 25 (mild disability), 50 (moderate), 75 (severe) and 100 (unable to perform activities). Higher scores indicate greater limitation.
Time Frame: At Baseline
Population: Only a subset of participants completed the questionnaire at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 12 | 13
score on a scale | 12.40 (16.83) | 21.45 (18.44)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.096, t-test, 2 sided

21. Secondary Outcome: Mean Disability of Arm, Shoulder, Hand Questionnaire (DASH) Scores
Description: as for outcome 20
Time Frame: At 4 weeks
Population: Only a subset of participants completed the questionnaire at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 12 | 13
score on a scale | 11.20 (16.03) | 17.62 (18.22)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.206, t-test, 2 sided

22. Secondary Outcome: Mean Patient-Reported Outcomes Measurement Information System® (PROMIS) Physical Function for the Upper Extremity (UE)
Description: The PROMIS for the Upper Extremity is reliable and addresses disability with physical activities that involve upper limb activities. The instrument items include 5 response options, from 1 "not at all" to 5 "very much." Total scores range from 0 to 100. PROMIS UE scores are scored using a T-score metric, with higher scores indicate higher levels of physical functioning of the upper extremity.
Time Frame: At Baseline
Population: Only a subset of participants completed the questionnaire at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 11 | 10
score on a scale | 47.86 (6.26) | 44.70 (7.71)

23. Secondary Outcome: Mean Patient-Reported Outcomes Measurement Information System® (PROMIS) Physical Function for the Upper Extremity (UE)
Description: as for outcome 22
Time Frame: At 4 weeks
Population: Only a subset of participants completed the questionnaire at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 11 | 10
score on a scale | 49.35 (6.40) | 43.14 (8.44)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.080, t-test, 2 sided

24. Secondary Outcome: Mean Scores on the Participant Version of the Patient-Reported Outcomes Measurement Information System (PROMIS®-29) (Version 2)
Description: The PROMIS 29 v2.0 profile assesses pain intensity using a response scale for each item ranging from 0 (no pain) to 10 (worst imaginable pain) on seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance), with four items per domain and one question which addresses pain intensity item. PROMIS-29 domains are scored using a T-score metric, with higher scores indicate higher levels of functioning.
Time Frame: At Baseline
Population: Only a subset of participants completed the questionnaire at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 11 | 10
score on a scale
  Physical Function | 19.4 (1.0) | 17.6 (2.6)
  Anxiety | 6.5 (3.0) | 6.8 (3.5)
  Depression | 5.7 (2.3) | 6.5 (3.5)
  Fatigue | 7.0 (2.7) | 9.6 (3.0)
  Sleep Disturbance | 8.6 (3.3) | 10.0 (2.2)
  Roles/Activity | 18.1 (2.3) | 15.1 (3.1)
  Pain Interference | 4.5 (1.5) | 7.5 (2.8)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Physical Function Domain; Test type: Other; p = 0.068, t-test, 2 sided
Statistical Analysis 2: Comparison: Manual Lymph Drainage vs Negative Pressure; Anxiety Domain; Test type: Other; p = 0.808, t-test, 2 sided
Statistical Analysis 3: Comparison: Manual Lymph Drainage vs Negative Pressure; Depression Domain; Test type: Other; p = 0.557, t-test, 2 sided
Statistical Analysis 4: Comparison: Manual Lymph Drainage vs Negative Pressure; Fatigue Domain; Test type: Other; p = 0.049, t-test, 2 sided
Statistical Analysis 5: Comparison: Manual Lymph Drainage vs Negative Pressure; Sleep Disturbance Domain; Test type: Other; p = 0.279, t-test, 2 sided
Statistical Analysis 6: Comparison: Manual Lymph Drainage vs Negative Pressure; Roles/Activity Domain; Test type: Other; p = 0.020, t-test, 2 sided
Statistical Analysis 7: Comparison: Manual Lymph Drainage vs Negative Pressure; Pain Interference Domain; Test type: Other; p = 0.009, t-test, 2 sided

25. Secondary Outcome: Mean Scores on the Participant Version of the Patient-Reported Outcomes Measurement Information System (PROMIS®-29) (Version 2)
Description: as for outcome 24
Time Frame: At 4 weeks
Population: Only a subset of participants completed the questionnaire at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 11 | 9
score on a scale
  Physical Function | 19.8 (0.40) | 17.2 (3.4)
  Anxiety | 4.9 (1.3) | 6.7 (3.0)
  Depression | 4.5 (1.0) | 5.1 (2.2)
  Fatigue | 6.5 (2.8) | 8.9 (3.2)
  Sleep Disturbance | 8.0 (3.1) | 10.4 (4.1)
  Roles/Activity | 18.5 (2.4) | 13.9 (3.9)
  Pain Interference | 4.9 (1.4) | 7.9 (4.0)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Physical Function Domain; Test type: Other; p = 0.038, t-test, 2 sided
Statistical Analysis 2: Comparison: Manual Lymph Drainage vs Negative Pressure; Anxiety Domain; Test type: Other; p = 0.108, t-test, 2 sided
Statistical Analysis 3: Comparison: Manual Lymph Drainage vs Negative Pressure; Depression Domain; Test type: Other; p = 0.467, t-test, 2 sided
Statistical Analysis 4: Comparison: Manual Lymph Drainage vs Negative Pressure; Fatigue Domain; Test type: Other; p = 0.078, t-test, 2 sided
Statistical Analysis 5: Comparison: Manual Lymph Drainage vs Negative Pressure; Sleep Disturbance Domain; Test type: Other; p = 0.147, t-test, 2 sided
Statistical Analysis 6: Comparison: Manual Lymph Drainage vs Negative Pressure; Roles/Activity Domain; Test type: Other; p = 0.004, t-test, 2 sided
Statistical Analysis 7: Comparison: Manual Lymph Drainage vs Negative Pressure; Pain Interference Domain; Test type: Other; p = 0.032, t-test, 2 sided

26. Secondary Outcome: Mean Functional Assessment of Cancer Therapy-Breast (FACT-B) Scores
Description: The FACT-B is a self-report instrument that measures multidimensional quality of life (QOL) in patients with breast cancer. The FACT-B consists of 37 questions that address physical, social, emotional, and functional well-being, with specific questions relevant to women with breast cancer. Each item has a score range of 0 (Not at all) to 4 (Very much), with a total score ranging from 0-148 The higher the score, the better the QOL reported by the participant.
Time Frame: At Baseline
Population: Only a subset of participants completed the questionnaire at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 12 | 14
score on a scale | 114.3 (21.8) | 113.6 (21.1)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.938, t-test, 2 sided

27. Secondary Outcome: Mean Functional Assessment of Cancer Therapy-Breast (FACT-B) Scores
Description: as for outcome 26
Time Frame: At 4 weeks
Population: Only a subset of participants completed the questionnaire at week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 12 | 14
score on a scale | 118.4 (14.4) | 114.7 (18.8)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.603, t-test, 2 sided

28. Secondary Outcome: Mean Body Image Scale (BIS) Score
Description: The 10-item Body Image Scale was developed by Hopwood et al. in 2001 to measure affective, behavioral, and cognitive body image symptoms. Patients can indicate body image symptoms on a 4-point scale (0 "not at all" to 3 "very much"). The total score ranges from 0 to 30 and can be calculated by summing up the 10 items. A higher score means a higher level of body image disturbance
Time Frame: At baseline
Population: Only a subset of participants completed the assessment at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 12 | 13
score on a scale | 8.8 (6.6) | 9.4 (8.4)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.837, t-test, 2 sided

29. Secondary Outcome: Mean Body Image Scale (BIS) Score
Description: as for outcome 28
Time Frame: At 4 weeks
Population: Only a subset of participants completed the questionnaire at week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 12 | 13
score on a scale | 7.7 (6.4) | 9.5 (7.5)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.511, t-test, 2 sided

30. Secondary Outcome: Mean Functional Assessment of Chronic Illness Therapy (FACIT) - Treatment Satisfaction - General (TSG) Scores
Description: Satisfaction with treatment will be evaluated at the 4-week assessment using the Functional Assessment of Chronic Illness Therapy (FACIT) - Treatment Satisfaction - General (TSG) (FACIT-TSG- Version 4). The FACIT-TSG is a copyrighted 8-item questionnaire, with each item score ranging from 0 ("not at all") to 4 ("very much"). Total scores range from 0 to 32 with higher scores indicating greater satisfaction with treatment.
Time Frame: At 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Manual Lymph Drainage | Negative Pressure
Number analyzed (Participants) | 12 | 10
score on a scale | 24.6 (5.9) | 27.0 (5.2)
Statistical Analysis 1: Comparison: Manual Lymph Drainage vs Negative Pressure; Test type: Other; p = 0.326, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Arm/Group | Manual Lymph Drainage | Negative Pressure
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 1/13 | 4/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Manual Lymph Drainage (N=13) | Negative Pressure (N=15)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Elbow Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Limb Pain (General disorders) | 0 (0) | 1 (1)
Shoulder/Neck Pain (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT03252145/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT03252145/Prot_SAP_001.pdf